CLINICAL TRIAL: NCT03465930
Title: Histologic Analysis of the Lymphatic Collecting Vessels Used for Minimally Invasive Supermicrosurgical Lymphatico-venous Anastomoses in the Treatment of Lymphedema
Brief Title: Histologic Analysis of the Lymphatic Vessels Used for Supermicrosurgical Lymphatico-venous Anastomoses in Lymphedema
Acronym: s-LVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paolo Gennaro (Other)
Collaborators: Elisabetta Weber, MD (Unknown)
Responsible Party: Sponsor-Investigator, Paolo Gennaro, MD, PhD. Associate Professor of Maxillofacial Surgery, University of Siena, University of Siena
Organization: University of Siena (Other)
Other Study IDs: LVA2017
Record Dates: First submitted 2017-12-07; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Lymphedema
Keywords: Lymphedema; Lymphatic collecting vessels; Supermicrosurgery; Lymphatic-venous anastomoses; Immunohistochemistry
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biospecimens to be retained are tissue, more precisely they are segments of the lymphatic vessels which are to be anastomosed with the veins, they are therefore very small structures (maximum 0.4mm diameter, 2-5mm in length) that are removed for technical reasons in a variable number between 1 and 3 for each patient during surgery. This doesn't affect in any way the success of the surgery itself. These samples instead of being destroyed, will be formalin fixed and transported to the laboratory of Prof. Elisabetta Weber where they will be paraffin embedded. Histologic sections will be obtained and adequate staining will be made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lymphedema: Patients affected by primary or secondary lymphedema. The intervention will consist in supermicrosurgical lymphatico-venous anastomoses (sLVA) to allow drainage of the lymph in the venous stream distal to the obstruction. sLVA is a minimally invasive procedure performed under local anesthesia. It requires an accurate visualization of the lymphatic vessels that are still functional.
  Interventions: Procedure: Supermicrosurgical lymphatico-venous anastomoses

INTERVENTIONS:
Procedure: Supermicrosurgical lymphatico-venous anastomoses — Supermicrosurgical lymphatico-venous anastomoses (sLVA) require an accurate visualization of the lymphatic vessels that are still functional. Lymphatic vessels are visualized with lymphography using a fluorescent dye, indocyanine green. Adjacent superficial veins mapping is obtained with Accuvein device.

SUMMARY:
Lymphedema, primary or secondary, is a chronic disease that causes functional impairment and has an important impact on patient's quality of life. Lymphedema can be primary or secondary. Secondary lymphedema, which is more common, especially in industrialized countries, is often due to surgery and radiotherapy to treat cancer. There is no definite cure for lymphedema; conservative treatments such as elastic compression garments, bandages and manual lymphatic drainage help reducing the edema but do not resolve it. Many types of surgery have been used in the past, the most recent are lymphatic-venous anastomoses, a minimally invasive procedure that may be performed under local anesthesia. Briefly, after visualizing the lymphatic vessels with a fluorescent dye, one or more anastomosis are created between collecting lymphatic vessels and superficial veins in order to drain the lymph into the blood stream bypassing the obstacle. During this procedure, it is possible to take samples of the collecting lymphatic vessels that are to be anastomosed with veins and use them for histological and immunohistochemical studies, without causing any additional discomfort to the patient. These samples can be formalin fixed and paraffin embedded. The obtained sections will be stained with a lymphatic endothelium marker and a smooth muscle specific stain. A morphometric study will be conducted and, based on the results a statistical evaluation will be made. The analysis will be conducted on samples obtained from patients, affected by secondary or primary lymphedema willing to provide their free and informed consent. The aim of this study is to evaluate the histopathological characteristics of the collecting lymphatic vessels that have been anastomosed with adjacent veins during surgery, and relate the results with the obtained clinical response. The acquired knowledge will contribute to optimize the clinical approach to prevent and treat lymphedema, by helping to select the patients that will benefit more from the surgery, and to select vessels and anatomical sites that have better chances to provide efficient anastomoses.

DETAILED DESCRIPTION:
Background:

Lymphedema is a chronic pathologic condition that causes significant functional impairment to the patient and has a great impact on his quality of life. It may be primary or secondary. Secondary lymphedema, that is the most common, is generally due to surgery and radiotherapy for cancer, particularly of the breast, uterus and prostate but can also occur after a trauma. Primary lymphedema can be congenital or begin at puberty, or more rarely after age 35, in this case, often following a trigger event such as trauma or infection.

There is no specific treatment for this highly disabling disease and patients must lifelong try to reduce edema and limit its progression by the use of elastic compression garments and with manual lymphatic drainage. Over the years several surgical approaches have been proposed, including more recently super microsurgical lymphatic-venous anastomosis (sLVA) to allow drainage of the lymph in the venous stream distal to the obstruction. sLVA is a minimally invasive procedure performed under local anesthesia with discharge the day after surgery. It requires an accurate visualization of the lymphatic vessels that are still functional. Lymphatic vessels are visualized with lymphography using a fluorescent dye, indocyanine green. In selected cases, magnetic resonance can also be useful. Small samples of the vessel selected to perform the LVA can easily be taken during surgery, formalin-fixed and paraffin-embedded for histologic and immunohistochemical studies without further discomfort or complications for the patient.

Knowledge on the histopathological aspects of lymphedema is extremely limited, this study must therefore be considered an exploratory one, possibly intended to generate more hypotheses than to solve them. A better understanding of the physio-pathological mechanisms of lymphedema can lead to a more effective surgical approach and, in selected cases, even prevent its development with considerable advantages in terms of the patient's quality of life and also in reducing national health care system costs (direct costs arising from the need to undergo continuous physiotherapy and indirect costs due to disability, serious intercurrent infections requiring hospitalization and loss of work days).

Primary purpose of the study is to evaluate the histopathologic features of the lymphatic vessels anastomosed with veins. The primary purpose will be divided in two phases: 1. on secondary lymphedema; 2. on primary lymphedema.

Secondary purpose of the study is the correlation of histopathologic parameters with other clinical data: type of lymphedema (primary versus secondary), age of the patient, years from the onset of the disease, anatomic site of the anastomosis, morphologic characteristics of the vessel as assessed pre-operatively by lymphography and or magnetic resonance imaging.

The acquired knowledge will be valuable to customize the approach to prevent and treat lymphedema. In particular, will help to:

1. Select patients who can better benefit from sLVA and within them prioritize intervention.
2. Select the lymphatic vessels that are more likely to give an efficient anastomosis with veins.
3. Based on the comparison between the morphological features of lymphatic vessels of various parts of the limb affected by lymphedema, select the anatomical sites where efficient anastomosis are more likely to be achieved.

Experimental design This is a single center, non commercial laboratory study to be performed on human biological material. Patients will be recruited with a consecutive participant sampling of all those who meet the eligibility criteria and are willing to provide informed consent. Samples of the lymphatic vessels to be anastomosed with veins will be taken at time of sLVA, this can be done without any inconvenience for the patient because the lymphatic vessels are often too long and a segment must be removed to perform the anastomosis. Usually during surgery 1-3 lymphatic vessels/patient are removed for technical reasons. These samples instead of being destroyed, will be transported to the laboratory of Prof. Elisabetta Weber where they will be formalin-fixed and paraffin embedded. Histologic and immunohistochemical studies will be performed on the obtained sections stained with appropriate markers and or/stains for the lymphatic endothelium (D2-40 and VEGFR-3) and of smooth muscle cells. Appropriate stains will be used to determine the relative proportions of smooth muscle cells and collagen fibers in the lymphatic wall. A morphometric analysis of data will be performed and data will be related with the clinical results obtained.

All data will be statistically evaluated. As there are no previous experiences that allow to estimate the variability of the parameters in the study, it is not possible to hazard a formal analysis of the statistical power of the study. However, a sample of 25 patients should be sufficient to provide a first estimate of the variability of the parameters and inform future efficacy studies based on the hypothesis testing model tests (Tukey, 1977). Since the sample comprises two different types of lymphedema, primary and secondary, a minimum of 25 patients is required to have a sufficient number of patients for each of these two groups. It will not be difficult to find cases of secondary lymphedema, since it is very common (especially in industrialized countries, as a consequence of surgery and radiotherapy for cancer treatment), while it will be more difficult to find cases of primary lymphedema since this type of lymphedema is rare and often undiagnosed or misdiagnosed. Should the individual variability be considerable, it would be necessary to increase the number of patients. Finally, it should be noted that, given the small size of the samples (maximum of 0.4mm diameter, 2-5mm in length), not all histological preparations will be successful. Therefore, the investigators believe it prudent to set a maximum number of samples of 200.

The statistical analysis will make use, as well as of descriptive methods, of methods of comparison and correlation of parametric (Student t, linear correlation) or non-parametric (logistics analysis, chi-square, Spearman's rank correlation), in agreement to the features of the data distribution that will be found. The correlation between the time from onset of lymphedema and primary and secondary outcomes will be investigated with Cox proportional hazard model. Differences in outcome measures between recent (<1 year) and long standing lymphedema will be investigated using Generalized Linear Models using gaussian family and identity link. When more than one sample from the same patient is present, the patient will be included in the model as a random effect variable. A p value of 0.05 or less for a two tails distribution will be considered statistically significant. Data is presented as M ± robust SE All the analyses will be performed using Stata vers. 12 (Stata Corp, College Station, TX).

Aim of the study:

The aim is to better understand the pathogenetic aspects and pathophysiology of lymphedema (of which very little is known) and evaluate the structure of lymphatic vessel in relation to the stage of lymphedema, to optimize the choice of the lymphatic vessels better suited to achieve functioning anastomoses. The obtained data will be correlated with clinical outcome which will be evaluated with the following objective parameters: reduction in limb circumference measured at several points (hand, wrist, -5 cm from the elbow, elbow and +5 cm from the elbow; for leg: foot, ankle, -10 cm from the knee, the knee, to +10 cm from the knee); reduction/absence of episodes of lymphangitis; decreasing compression class of elastic compression garments. Subjective parameters will also be evaluated as indexes of the patient's life quality: reduction of discomfort, reduced sense of heaviness, ability to wear clothes more easily, improved social life.

The study will be conducted in accordance with the ethical principles in the Declaration of Helsinki in its latest revision. Participation in the study will be subject to obtaining the free and informed consent.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old;
* patients affected by primary or secondary lymphedema;
* patients willing to give their free and informed consent.

Exclusion Criteria:

* patients currently undergoing radiotherapy;
* patients currently undergoing chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients affected by lymphedema that come to us to undergo s-LVA surgery, that match the eligibility criteria and give their free and informed consent. There is no restriction of sex, gender, race, ethnics, country, region, town, etc.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Expression of the lymphatic endothelial marker D2-40 in relation with the duration of lymphedema. | Collection of samples from different sites of at least 10 patients will require at least 6 months
  On sections stained with D2-40, under light microscopy with the aid of the morphometric program NIS elements tracing the portions of the endothelium stained positively for this marker and comparing the sum of all positive segments of each vessel with the length of its inner profile. The duration of lymphedema in number of years can be obtained using previous medical records (e.g. lymphography or lymphoscintigraphy) when the patient comes to observation after the diagnosis has already been made or, when no previous medical record is available, through the anamnesis. The duration of lymphedema from clinical onset to the time of surgery is expressed in number of years.

SECONDARY OUTCOMES:
Area of the vessel wall versus area of the lumen | Collection of samples from different sites of at least 10 patients will require at least 6 months
  Subtracting the inner from the outer profile with the aid of the morphometric program NIS elements.
The relative proportion of smooth muscle cells and collagen fibers in the lymphatic vessel wall. | Collection of samples from different sites of at least 10 patients will require at least 6 months
  Staining with Trichrome stain and measuring the threshold of the stained area (threshold of red for smooth muscle cells, threshold of blue for collagen fibers).
Differences in the histology of lymphatics between primary and secondary lymphedema. | Since primary lymphedema is rare, collection of an adequate number of cases of primary lymphedema (at least 10) to evaluate whether there are histologic differences with secondary lymphedema will require at least three years.
  Histologic measurements are the same as for the primary outcome. To determine if the lymphedema is primary or secondary an accurate anamnesis is usually enough: patients report history of trauma or cancer treatment in case of secondary lymphedema, no such events in primary lymphedema.
Relation between the anatomic site of the anastomosis and histologic parameters. | Collection of samples from different sites of at least 10 patients will require at least 6 months.
  Measurement of histologic parameters as in the primary outcome, comparison between samples taken from different sites of the same patient (hand or wrist versus elbow, or more rarely arm, for the upper limb, foot or ankle versus knee or more rarely thigh, for the lower limb).
Correlation between histologic modifications and morphologic appearance at lymphography and / or at MRL (Magnetic Resonance Lymphography). | Collection of samples from different sites of at least 10 patients will require at least 6 months
  Lymphography with a fluorescent dye (indocyanine green), routinely performed prior to surgery to choose the lymphatic vessels suitable for anastomoses. In later stage lymphedemas, MRL, with gadolinium as a contrast medium, is sometimes necessary to allow visualization of lymphatic vessels thanks to the slow wash out of gadolinium. Histologic evaluation as in the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gennaro, MD, PhD, Study Director — Department of Biotechnology, University of Siena; Department of Maxillofacial Surgery, Azienda Ospedaliera Universitaria Senese; Elisabetta Weber, MD, Principal Investigator — University of Siena, Dept. of Molecular and Developmental Medicine.
Locations (1):
- Dept. of Maxillofacial Surgery, Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided
For technical reasons we do not yet know which type of data may be obtained and hence cannot make plans for data sharing.

REFERENCES:
- [Background] Koshima I, Inagawa K, Urushibara K, Moriguchi T. Supermicrosurgical lymphaticovenular anastomosis for the treatment of lymphedema in the upper extremities. J Reconstr Microsurg. 2000 Aug;16(6):437-42. doi: 10.1055/s-2006-947150. PMID 10993089
- [Background] Yamamoto T, Narushima M, Yoshimatsu H, Seki Y, Yamamoto N, Oka A, Hara H, Koshima I. Minimally invasive lymphatic supermicrosurgery (MILS): indocyanine green lymphography-guided simultaneous multisite lymphaticovenular anastomoses via millimeter skin incisions. Ann Plast Surg. 2014 Jan;72(1):67-70. doi: 10.1097/SAP.0b013e3182605580. PMID 23241778
- [Background] Mihara M, Hara H, Hayashi Y, Narushima M, Yamamoto T, Todokoro T, Iida T, Sawamoto N, Araki J, Kikuchi K, Murai N, Okitsu T, Kisu I, Koshima I. Pathological steps of cancer-related lymphedema: histological changes in the collecting lymphatic vessels after lymphadenectomy. PLoS One. 2012;7(7):e41126. doi: 10.1371/journal.pone.0041126. Epub 2012 Jul 24. PMID 22911751
- [Background] Mihara M, Murai N, Hayashi Y, Hara H, Iida T, Narushima M, Todokoro T, Uchida G, Yamamoto T, Koshima I. Using indocyanine green fluorescent lymphography and lymphatic-venous anastomosis for cancer-related lymphedema. Ann Vasc Surg. 2012 Feb;26(2):278.e1-6. doi: 10.1016/j.avsg.2011.08.007. Epub 2011 Nov 12. PMID 22079465
- [Background] Liu NF, Lu Q, Liu PA, Wu XF, Wang BS. Comparison of radionuclide lymphoscintigraphy and dynamic magnetic resonance lymphangiography for investigating extremity lymphoedema. Br J Surg. 2010 Mar;97(3):359-65. doi: 10.1002/bjs.6893. PMID 20101589
- [Background] Yamamoto T, Yamamoto N, Yamashita M, Furuya M, Hayashi A, Koshima I. Efferent Lymphatic Vessel Anastomosis: Supermicrosurgical Efferent Lymphatic Vessel-to-Venous Anastomosis for the Prophylactic Treatment of Subclinical Lymphedema. Ann Plast Surg. 2016 Apr;76(4):424-7. doi: 10.1097/SAP.0000000000000381. PMID 25389716
- [Background] Kahn HJ, Marks A. A new monoclonal antibody, D2-40, for detection of lymphatic invasion in primary tumors. Lab Invest. 2002 Sep;82(9):1255-7. doi: 10.1097/01.lab.0000028824.03032.ab. No abstract available. PMID 12218087
- [Background] Nagase T, Gonda K, Inoue K, Higashino T, Fukuda N, Gorai K, Mihara M, Nakanishi M, Koshima I. Treatment of lymphedema with lymphaticovenular anastomoses. Int J Clin Oncol. 2005 Oct;10(5):304-10. doi: 10.1007/s10147-005-0518-5. PMID 16247656
- [Result] Gennaro P, Borghini A, Chisci G, Mazzei FG, Weber E, Tedone Clemente E, Guerrini S, Gentili F, Gabriele G, Ungari C, Mazzei MA. Could MRI visualize the invisible? An Italian single center study comparing magnetic resonance lymphography (MRL), super microsurgery and histology in the identification of lymphatic vessels. Eur Rev Med Pharmacol Sci. 2017 Feb;21(4):687-694. PMID 28272715
- [Result] Mihara M, Hara H, Kikuchi K, Yamamoto T, Iida T, Narushima M, Araki J, Murai N, Mitsui K, Gennaro P, Gabriele G, Koshima I. Scarless lymphatic venous anastomosis for latent and early-stage lymphoedema using indocyanine green lymphography and non-invasive instruments for visualising subcutaneous vein. J Plast Reconstr Aesthet Surg. 2012 Nov;65(11):1551-8. doi: 10.1016/j.bjps.2012.05.026. Epub 2012 Jul 19. PMID 22817883
- [Result] Mihara M, Hara H, Furniss D, Narushima M, Iida T, Kikuchi K, Ohtsu H, Gennaro P, Gabriele G, Murai N. Lymphaticovenular anastomosis to prevent cellulitis associated with lymphoedema. Br J Surg. 2014 Oct;101(11):1391-6. doi: 10.1002/bjs.9588. Epub 2014 Aug 13. PMID 25116167
- [Result] Gennaro P, Gabriele G, Mihara M, Kikuchi K, Salini C, Aboh I, Cascino F, Chisci G, Ungari C. Supramicrosurgical lymphatico-venular anastomosis (LVA) in treating lymphoedema: 36-months preliminary report. Eur Rev Med Pharmacol Sci. 2016 Nov;20(22):4642-4653. PMID 27906440

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT03465930/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT03465930/SAP_001.pdf